CLINICAL TRIAL: NCT06796998
Title: Phase 2 Trial of Epcoritamab in Patients With Newly Diagnosed Marginal Zone Lymphoma (MZL)
Brief Title: Epcoritamab in Patients With Newly Diagnosed Marginal Zone Lymphoma (MZL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Izidore Lossos, MD (Other)
Collaborators: Genmab (Industry); AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Izidore Lossos, MD, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240621; NCI-2025-06276 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Marginal Zone Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Splenic Marginal Zone Lymphoma; Nodal Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epcoritamab Group (Experimental): Participants will receive up to 12 cycles of Epcoritamab therapy, each cycle lasting 28 days.
  Total participation is up to 3 years.
  Interventions: Biological: Epcoritamab

INTERVENTIONS:
Biological: Epcoritamab — Epcoritamab will be administered via subcutaneous (SC) injection using a step-up dosing schedule as follows:
  * Cycle 1, Day 1: 0.16 mg
  * Cycle 1, Day 8: 0.8 mg
  * Cycle 1, Day 15: 3 mg
  * Cycle 1, Day 22: 48 mg
  * Cycles 2 to 3, Days 1, 8, 15 and 22: 48 mg
  * Cycles 4 to 9, Days 1 and 15: 48 mg
  * Cycles 10 to 12; Day 1: 48 mg

SUMMARY:
The purpose of this study is to assess if an investigational treatment of Epcoritamab will be beneficial for patients with Marginal Zone Lymphoma (MZL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or older at the time of signing informed consent.
2. Able and willing to sign the informed consent form (ICF).
3. Ability to comply with the trial protocol.
4. Histologically confirmed Marginal Zone Lymphoma (MZL) of Extranodal Marginal Zone Lymphoma (EMZL), Nodal Marginal Zone Lymphoma (NMZL) and Splenic Marginal Zone Lymphoma (SMZL) subtypes presenting with stage I-IV disease.
5. Previously untreated participants.

   1. Participants with H. pylori-positive gastric EMZL who received an initial treatment with currently accepted antibiotics may be considered eligible if, after antibiotic regimen, participant has histologically confirmed MZL.
   2. Participants who were previously treated with localized therapy (eg, radiation or surgery) and never received systemic therapy and present with recurrent disease are eligible upon histological confirmation of MZL.
6. Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥1 lesion that measures >1.5 cm in the longest diameter (LDi) and ≥1.0 cm in the longest perpendicular diameter as assessed by PET/CT, CT or MRI, especially in extranodal sites, per response criteria for lymphomas (Cheson, et al., 2014). Imaging must be conducted within 6 weeks prior to the start of therapy.

   1. Participants with skin EMZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that skin lesion measures ≥1.5 cm in diameter by tape measure and is documented by photo or there are ≥2 skin lesions measuring >1 cm in diameter on the body that cannot be incorporated in one radiation field and at least one of them is histologically confirmed as MZL.
   2. Participants with gastric EMZL histologically confirmed and need therapy but do not have measurable disease and in which response to treatment can be assessed by multiple random gastric biopsies per Groupe d'Etude des Lymphomes de l'Adult (GELA) criteria (Ruskoné Fourmestraux, et al., 2011).
   3. Participants with conjunctival EMZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that conjunctival lesion measures ≥1 cm in diameter by tape measure and is documented by photo or there are multiple conjunctival lesions measuring together >1.5 cm that cannot be treated by radiation because of previous radiation therapy, contraindications to radiation and patient refusal to receive radiation therapy. At least one of these lesions needs to be histologically confirmed as MZL.
   4. Participants with splenic MZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that bone marrow (BM) infiltration of MZL is histologically confirmed.
7. Participants will be asked to provide a lymph node or tissue biopsy from the most recent available archival tissue or undergo an incisional or excisional lymph node or tissue biopsy but this is not an exclusion criteria.

   a. Participants with splenic MZL who do not have a tumor to biopsy or an archival tumor tissue sample are eligible for participation provided participant is willing to undergo a BM biopsy or provide an archival BM biopsy that was obtained before the date of the first dose of study treatment; BM sample must show histologically confirmed infiltration of MZL
8. Participant should have at least one of the following criteria for treatment initiation:

   * Threatened extranodal organ function, especially for extranodal MZL
   * Involvement of ≥3 nodal sites, each with diameter of ≥3 cm
   * Any nodal or extranodal tumor mass with a diameter of ≥5 cm
   * B symptoms (fever ≥38 degrees Celsius of unclear etiology, night sweats, weight loss >10% within the prior 6 months) or other symptoms attributed to disease or specific organ involvement.
   * Risk of local compressive symptoms that may result in organ compromise
   * Splenomegaly >13 cm or splenic lesion without splenomegaly and needs treatments (e.g., symptoms, cytopenias [hemoglobin (HgB) <10 g/dL and platelet count ≤ 80 × 10^9 platelets/L attributable to lymphoma bone marrow infiltration, splenomegaly or autoimmunity], >5,000 lymphoma cells/mm3).
   * Threatened organ function, especially for extranodal MZL
   * Leukopenia attributed to MZL (leukocytes <1,000 cells/mm3)
   * Leukemia (>5,000 lymphoma cells/mm3)
   * Requirement for transfusion or growth factor support attributed to lymphoma
   * Involvement of 2 or more extranodal sites, with tumor/lesion in each extranodal site ≥1 cm
9. Life expectancy >3 months.
10. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
11. Adequate hematologic, hepatic, and renal function tested within 6 weeks prior to the start of therapy (values must not be achieved with growth factors):

    1. Absolute neutrophil count (ANC) ≥1.0 × 10^9 cells/L.
    2. Hemoglobin ≥8.0 g/dL.
    3. Platelet count ≥50 × 10^9 platelets/L.
    4. Total bilirubin ≤1.5 × upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin or lymphoma involvement of the liver and total bilirubin if ≤5 x ULN.
    5. Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤3.0 × ULN or ≤5 × ULN in the presence of liver involvement by lymphoma.
    6. Creatinine within normal institutional limits, or

       * calculated creatinine clearance ≥35 mL/min by the Cockcroft-Gault Equation (Cockcroft, 1976)
       * estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 using the Modification of Diet in Renal Disease formula for participants with creatinine levels above institutional normal (unless due to lymphoma)
12. Willingness to avoid pregnancy during the trial and for at least 90 days after the last dose of the trial intervention. For more information on Contraception, please see Section 5.12.

Exclusion Criteria:

1. Evidence of DLBCL transformation. Participants with presumptive evidence of transformation based on clinical assessment of factors such as, but not limited to, increasing lactate dehydrogenase (LDH), rapidly worsening disease, or frequent B-symptoms, must be ruled out for a transformation to a more aggressive disease, such as DLBCL.
2. History of central nervous system lymphoma (either primary or metastatic) or leptomeningeal disease. Participants with dural MZL are eligible.
3. Concurrent or previous anticancer therapy (eg, chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, investigational therapy, or tumor embolization).
4. Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone (>20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1.

   1. Steroids that are used for treatment of allergy or other underlying condition are permissible, but not steroids started to treat lymphoma. Participants receiving corticosteroids must be at a dose level ≤20 mg/day within 7 days of the trial intervention administration.
   2. The use of inhaled corticosteroids is permitted
   3. The use of mineralocorticoids for management of orthostatic hypotension is permitted
   4. Single dose of dexamethasone for nausea or B symptoms is permitted
   5. Antibiotic treatment of H. pylori-positive gastric EMZL
5. Allogeneic stem cell transplant or autologous stem cell transplant or chimeric antigen receptor (CAR) T-cell therapy for any indication
6. Active graft versus host disease.
7. Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
8. Current or previous other malignancy within 3 years of trial entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
9. Significant concurrent, uncontrolled medical condition, including, but not limited to, renal, hepatic, hematological, gastrointestinal (GI), endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
10. Chronic or current active infectious disease (including severe acute respiratory syndrome coronavirus (CoV) 2 (SARS-CoV-2)) requiring systemic antibiotics, antifungal, or antiviral treatment or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1.
11. Exposure to a live vaccine within 30 days of administration or anticipation that a live attenuated vaccine will be required during the study.

    1. Inactivated influenza vaccinations may be given during the influenza season.
    2. An approved coronavirus disease 2019 (COVID-19) vaccine (messenger ribonucleic acid (mRNA), inactivated virus, and replication deficient viral vector vaccines) is allowed.
12. Known human immunodeficiency virus (HIV) infection or positivity on immunoassay. Note: HIV screening test is optional
13. History of solid organ transplantation
14. History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies (Mabs)
15. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells or any component of the epcoritamab, lenalidomide, or thalidomide formulation, including mannitol.
16. Significant cardiovascular disease (eg, New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 3 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
17. Known or suspected chronic active Epstein-Barr virus (EBV) infection
18. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
19. History of progressive multifocal leukoencephalopathy (PML)
20. Active hepatitis B infection

    a. Patients who are hepatitis B surface antigen (HbsAg) negative and hepatitis B core antibody (HbcAb) positive must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation. Hepatitis B DNA must be negative prior to treatment with epcoritamab. Patients with chronic HBV infection who are at risk of viral reactivation (HBsAg positive and/or anti-hepatitis B core (anti-HBc) positive) must receive antiviral prophylaxis with nucleos(t)ide analogue with high barrier to resistance (tenofovir disoproxil fumarate, tenofovir alafenamide, or entecavir) as described in Section 7.2.4.5.
21. Active hepatitis C infection

    a. Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
22. History of autoimmune disease, including, but not limited to, myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

    1. Patients with a remote history of, or well-controlled, autoimmune disease with a treatment free interval from immunosuppressive therapy for 12 months may be eligible to enroll if judged to be safe by the Investigator
    2. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible
    3. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    4. Patients with a history of disease-related immune thrombocytopenic purpura, or autoimmune hemolytic anemia may be eligible
    5. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (eg, patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

       * i. Rash must cover 10% of body surface area
       * ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids
       * iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency oral corticosteroids within the previous 12 months
23. Patient has no known active SARS-CoV-2 infection. If a patient has signs/symptoms suggestive of SARS-CoV-2 infection, the patient must have a negative molecular (e.g., PCR) test or 2 negative antigen test results at least 24 hours apart.

    Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations. Patients who do not meet SARS-CoV-2 infection eligibility criteria must be screen-failed and may only rescreen if the following have been met:
    * At least 10 days since first positive test result have passed in asymptomatic patients or at least 10 days since recovery, defined as resolution of fever without use of antipyretics and improvement in symptoms.
24. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | 12 months
  The proportion of participants achieving a best overall response of complete response (CR) after Cycle 12 of study therapy will be reported. Response will be assessed using modified Cheson criteria, if disease is not fluorodeoxyglucose (FDG)-avid in initial Screening; or by revised Lugano criteria if Screening FDG-positron emission tomography (PET)/ computed tomography (CT) demonstrated FDG avid disease. For Lugano criteria, CR will be defined by a Deauville score of ≤3.

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 7 months
  The proportion of participants achieving a best overall response of complete response (CR) after Cycle 3 and Cycle 7 of study therapy will be reported. Response will be assessed using modified Cheson criteria, if disease is not fluorodeoxyglucose (FDG)-avid in initial Screening; or by revised Lugano criteria if Screening FDG-positron emission tomography (PET)/ computed tomography (CT) demonstrated FDG avid disease. For Lugano criteria, CR will be defined by a Deauville score of ≤3.
Partial Response (PR) | Up to 12 months
  The proportion of participants achieving a best overall response of partial response (PR) after Cycle 12 of study therapy will be reported. Response will be assessed using modified Cheson criteria or revised Lugano criteria (based on FDG avidity), among evaluable participants.
Complete Response | 24 months
  The proportion of participants achieving a best overall response of complete response (CR) at 24 months after initiation of treatment will be reported. Response will be assessed using modified Cheson criteria or revised Lugano criteria (based on FDG avidity), among evaluable participants.
Overall Response Rate (ORR) | Up to 12 months
  The proportion of participants achieving a best overall response of complete response (CR) or partial response (PR) after Cycles 3, Cycle 7, and Cycle 12 of study therapy will be reported. Response will be assessed per Cheson or revised Lugano criteria (based on FDG avidity) modified for marginal zone lymphoma (MZL), among evaluable participants.
Time to Response (TTR) | Up to 12 months
  The time to response (TTR) to treatment among participants will be reported. TTR is the time in months from Cycle 1 Day 1 to achievement of complete response (CR) or partial response (PR) after initiation of treatment.
Duration of Response (DOR) | Up to 36 months
  The duration of response (DOR) to treatment among participants will be reported. DOR is the time in months from achievement of complete (CR) or partial response (PR) to progression, relapse, or death. For event-free participants, follow-up will be censored at the last date of documented still on PR or CR.
Number of Participants Experiencing Treatment-Related Adverse Events | Up to 13 months
  The number of participants experiencing treatment-related adverse events/toxicity will be reported. Adverse events (AEs), including serious adverse events, will be assessed using the using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events (AEs) will be assessed during treatment and 30 (±7) days after the last dose of the trial intervention.
Number of Participants Experiencing Treatment-Related Serious Adverse Events (SAEs) | Up to 13 months
  Number of Participants Experiencing Treatment-Related Serious Adverse Events will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of Participants Experiencing Treatment-Related Cytokine Release Syndrome (CRS) Adverse Events | Up to 13 months
  The number of participants experiencing treatment-related Cytokine Release Syndrome (CRS) adverse events will be reported. CRS-related adverse events will be assessed using American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading Criteria.
Number of Participants Experiencing Treatment-Related Clinical Tumor Lysis Syndrome (CTLS) Adverse Events | Up to 13 months
  The number of participants experiencing treatment-related clinical tumor lysis syndrome (CTLS) adverse events will be reported. CTLS-related adverse events will be assessed using Cairo-Bishop criteria.
Number of Participants Experiencing Treatment-Related Immune effector Cell-associated Neurotoxicity Syndrome (ICANS) Adverse Events | Up to 13 months
  The number of participants experiencing treatment-related immune effector cell-associated neurotoxicity syndrome (ICANS) adverse events will be reported. ICANS-related adverse events will be assessed using Lee et al., 2019 criteria.
Progression-Free Survival (PFS) | Up to 36 months
  Progression- Free Survival (PFS) among participants will be reported. PFS is defined as the elapsed time in months from start of treatment to documented progressive disease or death from any cause. For participants alive and progression-free, follow-up will be censored at the last date of documented progression-free status.
Overall Survival (OS) | Up to 36 months
  Overall Survival (OS) among participants will be reported. OS is defined as the elapsed time in months from start of treatment to death from any cause. Alive participants will be censored at last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Izidore Lossos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No